CLINICAL TRIAL: NCT02408393
Title: MIRs03: A Double-blind Randomized Trial of Paravertebral Block With Ropivacaine Before Breast Cancer Surgery: Effects on Chronic Postoperative Pain
Brief Title: MIRs03: Paravertebral Block With Ropivacaine Before Breast Cancer Surgery
Acronym: MIRs03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC 2014-07
Record Dates: First submitted 2015-03-17; First posted 2015-04-03 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Malignant Neoplasm of Breast
Keywords: Surgery; Paravertebral block; Chronic pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline (30 mL maximum)
  Interventions: Drug: Saline
- Ropivacaine (Experimental): Ropivacaine 7.5 mg/mL (0.35 mL/kg of solution)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Saline
  Other Names: NA Cl 0.9%
  Arms: Placebo
Drug: Ropivacaine
  Other Names: Naropeine
  Arms: Ropivacaine

SUMMARY:
Compare the effect of paravertebral block (PVB) with Ropivacaine or placebo on the incidence of chronic pain 3 months after breast cancer surgery.

DETAILED DESCRIPTION:
Before anesthesia, the second or third intercostal space is located. After an aspiration, 0.35 mL/kg of solution (ropivacaine 7.5 mg/mL or saline, maximum 30 mL) are injected into the paravertebral space. After 30 minutes, spread of PVB is evaluated by cold test on skin. Then, general anesthesia is induced.

Evaluation of the frequency of chronic pain at 3, 6 and 12 months by the Brief Pain Inventory (BPI) questionnaire and Neuropathic Pain Diagnostic (DN4) and Anxiety and depression evaluation by the Hospital Anxiety and Depression questionnaire (HAD) will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Women with non-metastatic invasive breast carcinoma or breast carcinoma in situ treated by:

   * either breast-conserving surgery with axillary lymph node dissection
   * either radical surgery with or without axillary lymph node dissection.
2. 18 years ≤ Age ≥ 85 years.
3. ASA class 1, 2 or 3.
4. No analgesic treatment for 2 days (no pre-existing chronic pain)
5. If a biological control has been requested recently or deemed necessary by the Investigator, then it should be satisfactory : Adequate hematologic and hemostasis: neutrophil count (ANC) > 1500/mm3, haemoglobin > 9 g/dl and platelets > 75 000/mm3, prothrombin time > 70%, activated partial thromboplastin time < 1.5 X Upper Limit of Normal (ULN)
6. Life expectancy ≥ 2 years.
7. Signed informed consent form.
8. Patient able to meet the self-assessments questionnaires (sufficient understanding assessments, proficiency in French)
9. Patient affiliated with a health insurance scheme (beneficiary or legal)

There is no prohibition for people to take part simultaneously in another search and there is no exclusion cause at the end of the research period.

Exclusion Criteria:

1. Ongoing neoplasm or history of malignancy other than breast cancer with the exception of: basal cell carcinoma, cervical carcinoma in situ, other treated cancer that has not relapsed during the 5 years preceding inclusion in the trial.
2. Bilateral breast carcinoma at the inclusion
3. Male subjects.
4. Metastatic breast carcinoma at diagnosis (M1).
5. Severe heart, liver and respiratory failure (ASA 4)
6. Allergy to local anesthetics and morphine.
7. Use of analgesics during the 48 hours preceding the surgical procedure.
8. History of breast surgery with painful sequelae
9. Major deformation of the spine
10. Puncture site infection
11. History of substance abuse.
12. Pregnant or lactating women, or women of childbearing potential without effective contraception
13. Subjects deprived of their liberty or under guardianship (including temporary guardianship).
14. Subjects unable to comply with medical follow-up of the trial for geographical, social or psychological reasons.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
To compare chronic pain 3 months after breast surgery in each arm | 3 months
  Percentage of patients who reported chronic pain 3 months after breast surgery in each arm evaluated by the Brief Pain Inventory, French version. Chronic pain is defined by the item 5 of BPI (upper or equal to 3)

SECONDARY OUTCOMES:
To measure the extend of dermatomes blocked | one year after surgery
  The extent of dermatomes blocked as measured by clinical examination to determine area where temperature perception change
To measure acute postoperative pain (Visual Analog Scale (VAS) | 48 postoperative hours
  Patient satisfaction on Visual Analog Scale (VAS)
To determine analgesic consumption | 48 postoperative hours
  consumption during the first 48 postoperative hours: morphine paracetamol and ketoprofen
To examine incidence of nausea and vomiting | 48 postoperative hours
  Common Toxicity Criteria for Adverse Effects (CTCAE) V4.03
To characterize chronic pain (Neuropathic Pain Diagnostic DN4 Questionnaire) | 3 months
  Neuropathic Pain Diagnostic DN4 Questionnaire
To evaluate the frequency of chronic pain (BPI questionnaire and Neuropathic Pain Diagnostic (DN4) | 6 and 12 months
  BPI questionnaire and Neuropathic Pain Diagnostic (DN4)
To compare presence of lymphedema | 3, 6 and 12 months
  Clinical examination
To evaluate anxiety and depression evaluation (Hospital Anxiety and Depression questionnaire (HAD) | 3, 6 and 12 months
  Hospital Anxiety and Depression questionnaire (HAD)
To evaluate complications of paravertebral block (CTCAE V4.03) | 12 months
  CTCAE V4.03
To determine the number of patients reporting pain at 6 months | 6 months
  Clinical examination to confirm the results of Visual analog scale, pain scores BPI and DN4

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FUMOLEAU, PHD, Study Director — drci.promotion@curie.fr
Locations (6):
- France (6):
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Centre Antoine LACASSAGNE, Nice
  - INSTITUT CURIE - Site Paris, Paris
  - Institut Curie site Saint-Cloud, Saint-Cloud
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cohen SP, Raja SN. Prevention of chronic postsurgical pain: the ongoing search for the holy grail of anesthesiology. Anesthesiology. 2013 Feb;118(2):241-3. doi: 10.1097/ALN.0b013e31827d4129. No abstract available. PMID 23340346
- [Result] Albi-Feldzer A, Mouret-Fourme E E, Hamouda S, Motamed C, Dubois PY, Jouanneau L, Jayr C. A double-blind randomized trial of wound and intercostal space infiltration with ropivacaine during breast cancer surgery: effects on chronic postoperative pain. Anesthesiology. 2013 Feb;118(2):318-26. doi: 10.1097/ALN.0b013e31827d88d8. PMID 23340351
- [Result] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Result] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Result] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770